CLINICAL TRIAL: NCT06170138
Title: An Explorative, Open-label, Randomised, 3-way Cross-over Study to Assess the Pharmacokinetics, Pharmacodynamics, Nicotine Extraction, Palatability, and Subjective Effects After Single Use of Nicotine Pouches in Daily Nicotine Users.
Brief Title: Study to Assess PK, PD, Nicotine Extraction, Palatability, Subjective Effects of Nicotine Pouches - Daily Nicotine Users
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amplicon AB (Industry)
Responsible Party: Sponsor
Organization: Emplicure AB (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AMP-01-101
Record Dates: First submitted 2023-11-23; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Nicotine Use Disorder
Keywords: nicotine; nicotine pouch products
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Each subject will be randomised to 1 of 6 IP use sequences The IPs will be administered as single pouches in a pre-determined randomised order.
  Test product 1 - Ampli-01 3 mg, nicotine pouch Test product 2 - Ampli-01 6 mg, nicotine pouch Comparator product - ZYN Cool Mint Mini Dry 6 mg nicotine /pouch Single 30-minutes IP use on 3 occasions (Visits 2 to 4).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ampli-01, 3 mg, nicotine pouch (Experimental): Subjects will report to the study site for a screening visit followed by 3 visits with a single IP use (Visits 2 to 4) on separate days.There will be at least 1 day between Visits 2, 3 and 4, respectively, where the subjects are allowed ad libitum use of their own nicotine product of choice. Each visit will last one day.
  Interventions: Other: Test product 1 - Test product 2 - Comparator product
- Ampli-01, 6 mg, nicotine pouch (Experimental): Subjects will report to the study site for a screening visit followed by 3 visits with a single IP use (Visits 2 to 4) on separate days.There will be at least 1 day between Visits 2, 3 and 4, respectively, where the subjects are allowed ad libitum use of their own nicotine product of choice. Each visit will last one day.
  Interventions: Other: Test product 1 - Test product 2 - Comparator product
- ZYN Cool Mint Mini Dry, 6 mg nicotine /pouch (Active Comparator): Subjects will report to the study site for a screening visit followed by 3 visits with a single IP use (Visits 2 to 4) on separate days.There will be at least 1 day between Visits 2, 3 and 4, respectively, where the subjects are allowed ad libitum use of their own nicotine product of choice. Each visit will last one day.
  Interventions: Other: Test product 1 - Test product 2 - Comparator product

INTERVENTIONS:
Other: Test product 1 - Test product 2 - Comparator product — Each subject will be randomised to 1 of 6 IP use sequences The IPs will be administered as single pouches in a pre-determined randomised order.
  Test product 1 - Ampli-01 3 mg, nicotine pouch Test product 2 - Ampli-01 6 mg, nicotine pouch Comparator product - ZYN Cool Mint Mini Dry 6 mg nicotine /pouch Single 30-minutes IP use on 3 occasions (Visits 2 to 4).

SUMMARY:
This is an explorative, open-label, randomised, 3-way cross-over study to assess pharmacokinetics (PK), pharmacodynamics (PD), safety and tolerability, nicotine extraction, palatability and subjective effects after single use of nicotine pouches in daily nicotine users.

DETAILED DESCRIPTION:
This is an explorative, open-label, randomised, 3-way cross-over, single use study, designed to assess the nicotine exposure from new nicotine pouch products.

A cross-over design was chosen to yield a more efficient comparison of the IPs than a parallel study design, i.e., fewer subjects are required since each subject will serve as its own control. To avoid carryover effects, subjects will abstain from oral tobacco/nicotine products as well as smoking (cigarettes or e-cigarettes) for at least 12 hours prior to each IP use (Visit 2-4).

Randomisation will be used to minimise bias in the assignment of subjects to an IP administration sequence and to increase the likelihood that known and unknown subject attributes (e.g., demographic and baseline characteristics) are evenly balanced.

The main purpose of this study is to understand the PK as well as to analyse the nicotine content left in pouch after use of Ampli01 and compare with a reference product. This will give consumers a better understanding of the behaviour of the product with the aim to be a potential satisfactory alternative to cigarette smoking. In addition, the safety profile, PD and subjective effects will be investigated and evaluated.

In summary, this study will provide critical data to assess PK, safety and formulation optimization to be able to provide consumers with a high-quality product. In addition, this study will contribute to the overall knowledge about nicotine pouches that can be of scientific value to improve public health strategies and regulations.

The study will include 12 randomised and evaluable subjects. The subjects are healthy male or female oral tobacco/nicotine pouch users aged 25 to 55 years, inclusive, who have used oral tobacco/nicotine products for ≥1 year, with a minimum daily consumption of 5 or more pouches (pouch strength 3-9 mg/pouch). Each subject will participate in the study for up to approximately 6 weeks, including the up to 28-day screening period.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Subjects who have used oral tobacco/nicotine products for ≥1 year, with a minimum daily consumption of 5 or more pouches with a pouch strength of 3-9 mg nicotine/pouch. Concomitant occasional use of other nicotine products (e.g., smoking, vaping) is allowed, as judged by the Investigator at the time of the screening visit.
3. Healthy male or female subject aged 25 to 55 years, inclusive, at the time of the screening visit.

   Female subjects of childbearing potential must be willing to use a sufficient contraceptive method for the duration of the study, this includes mechanical barrier (e.g., a male condom or a female diaphragm), combined [oestrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen-only hormonal anticonception associated with inhibition of ovulation [oral, injectable, implantable], intra uterine device (IUD) or intra uterine system (IUS). Sexual abstinence is allowed when this is the preferred and usual lifestyle of the subject.
4. Body Mass Index (BMI) ≥ 18.5 and ≤ 32.0 kg/m2 and a minimum weight of ≥ 50 kg.
5. Medically healthy subject without abnormal clinically significant medical history, physical findings, vital signs, ECG and laboratory values at the time of the screening visit, as judged by the Investigator.
6. Positive urine cotinine test (≥200 ng/mL) at the screening visit.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. After 10 minutes supine rest at the screening visit, any vital signs values outside the following ranges: - Systolic blood pressure: <90 or >140 mmHg, or - Diastolic blood pressure <50 or >90 mmHg, or - Pulse <40 or >90 bpm
3. Any surgical or medical condition, including abnormal salivation (also pharmaceutically induced), or history thereof, which, in the judgment of the Investigator, might interfere with the absorption, distribution, metabolism or excretion of the IP or may either put the subject at risk because of participation in the study, influence the results, or the subject's ability to participate in the study.
4. A history of diagnosed severe allergy/hypersensitivity or ongoing manifestations of severe allergy/hypersensitivity to aroma compounds (including fragrances and/or flavourings), as judged by the Investigator.
5. Any planned major surgery within the duration of the study.
6. Subjects who are pregnant, currently breastfeeding, or intend to become pregnant during the course of the study.
7. Any positive result at the screening visit for serum hepatitis B surface antigen, hepatitis C antibodies and/or HIV.
8. Positive screening result for drugs of abuse or alcohol at the screening visit or on admission to the study site prior to IP use at Visits 2 to 4. (Positive results that are expected given the subject's medical history and prescribed medications can be disregarded as judged by the Investigator.)
9. Presence or history of drug abuse, as judged by the Investigator.
10. History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
11. History of, or current use of anabolic steroids, as judged by the Investigator.
12. Current, ongoing use of beta-adrenergic blocking agents (beta blockers), including pro re nata (as needed) use.
13. Current, ongoing use of any medication known to be able to interfere with adrenaline testing, including but not limited to central nervous system stimulants (amphetamines), also including pro re nata (as needed) use, as judged by the Investigator.
14. Plasma donation within 1 month of the screening visit or blood donation (or corresponding blood loss) during the last 3 months prior to the screening visit.
15. Subjects who intend to change their nicotine consumption habit, including the intention to stop using nicotine products, within the next 3 months from the screening visit, as judged by the Investigator.
16. The Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2023-12-14 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
AUC from timepoint 0 to infinity (AUCinf), | Visit 2-4 (1 visit = 1 day): Pre-use and at 5, 10, 15, 20, 30, 40, 50, 60 minutes, 1 hour and 30 minutes, 2, 4, 6 and 8 hours post-IP use on visit 2, 3 and 4.
  Non-adjusted and baseline-adjusted PK parameters for nicotine including area under the curve (AUC) from timepoint 0 to infinity (AUCinf).
AUC from timepoint 0 to timepoint t (AUC0-t) | Visit 2-4 (1 visit = 1 day): Pre-use and at 5, 10, 15, 20, 30, 40, 50, 60 minutes, 1 hour and 30 minutes, 2, 4, 6 and 8 hours post-IP use on visit 2, 3 and 4.
  Non-adjusted and baseline-adjusted PK parameters for nicotine including AUC from timepoint 0 to timepoint t (AUC0-t).
AUC from timepoint 0 to 30 minutes (AUC0-30min) | Visit 2-4 (1 visit = 1 day): Pre-use and at 5, 10, 15, 20, 30, 40, 50, 60 minutes, 1 hour and 30 minutes, 2, 4, 6 and 8 hours post-IP use on visit 2, 3 and 4.
  Non-adjusted and baseline-adjusted PK parameters for nicotine including AUC from timepoint 0 to 30 minutes (AUC0-30min).
AUC from timepoint 0 to 60 minutes (AUC0-60min) | Visit 2-4 (1 visit = 1 day): Pre-use and at 5, 10, 15, 20, 30, 40, 50, 60 minutes, 1 hour and 30 minutes, 2, 4, 6 and 8 hours post-IP use on visit 2, 3 and 4.
  Non-adjusted and baseline-adjusted PK parameters for nicotine including AUC from timepoint 0 to 60 minutes (AUC0-60min).
Maximum plasma concentration (Cmax) | Visit 2-4 (1 visit = 1 day): Pre-use and at 5, 10, 15, 20, 30, 40, 50, 60 minutes, 1 hour and 30 minutes, 2, 4, 6 and 8 hours post-IP use on visit 2, 3 and 4.
  Non-adjusted and baseline-adjusted PK parameters for nicotine including maximum plasma concentration (Cmax).
Time to Cmax (Tmax) | Visit 2-4 (1 visit = 1 day): Pre-use and at 5, 10, 15, 20, 30, 40, 50, 60 minutes, 1 hour and 30 minutes, 2, 4, 6 and 8 hours post-IP use on visit 2, 3 and 4.
  Non-adjusted and baseline-adjusted PK parameters for nicotine including time to Cmax (Tmax).
Terminal elimination half-life (T1/2) | Visit 2-4 (1 visit = 1 day): Pre-use and at 5, 10, 15, 20, 30, 40, 50, 60 minutes, 1 hour and 30 minutes, 2, 4, 6 and 8 hours post-IP use on visit 2, 3 and 4.
  Non-adjusted and baseline-adjusted PK parameters for nicotine including terminal elimination half-life (T1/2).

SECONDARY OUTCOMES:
In vivo extracted amount (mg/unit) of nicotine | Visit 2-4 (1 visit = 1 day).
  In vivo extracted amount (mg/unit) of nicotine, for each investigational product (IP).
In vivo extracted fraction (%) of nicotine | Visit 2-4 (1 visit = 1 day).
  In vivo extracted fraction (%) of nicotine, for each investigational product (IP).
Highest recorded increase (Emax) in pulse rate from baseline. | Visit 2-4 (1 visit = 1 day): Pre-use and at 5, 10, 15, 20, 30, 40, 50, 60 minutes, 1 hour and 30 minutes, 2, 4, 6 and 8 hours post-IP use on visit 2, 3 and 4.
  Highest recorded increase (Emax) in pulse rate from baseline. Change from baseline.
Mean score for each palatability question 30 minutes after start of IP use. | Visit 2-4 (1 visit = 1 day): 30 minutes post-IP use on visit 2, 3 and 4.
  Mean score for each palatability question 30 minutes after start of IP use.
Urge-to-use | Visit 2-4 (1 visit = 1 day) : Pre-use and at 30, 60 minutes and 2 hours, post-IP use on visit 2, 3 and 4.
  Urge-to-use, product-liking, intent-to-use-again and onset-of-effect 30 minutes after start of IP use. Change from baseline for urge-to-use 30 minutes, 1 hour and 2 hours after start of IP use.
Adverse events (AEs). | Visit 2-4:All AEs (including SAEs) will be collected from the start of the first IP use until the last visit.
  Frequency, seriousness and intensity of adverse events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Erik Rein-Hedin, MD, Principal Investigator — Clinical Trial Consultants AB (CTC)
Locations (1):
- Clinical Trial Consultants AB (CTC), Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No